CLINICAL TRIAL: NCT03346239
Title: Effect of Attention Training or SSRIs on Symptoms and Neural Activation in Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Sheba Medical Center (Other Government); Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAUgcMRT
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Escitalopram; Dexetimide; Waiting Lists

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gaze Contingent Music Reward Therapy (Experimental): Participants will receive gaze-contingent feedback according to their viewing patterns, over a course of 12 weeks.
  Interventions: Behavioral: Gaze Contingent Music Reward Therapy
- Selective Serotonin Reuptake Inhibitors (Active Comparator): Participants will receive 10-20 mg of Escitalopram over a course of 12 weeks.
  Interventions: Drug: Escitalopram
- Waitlist Control (Placebo Comparator): Participants will wait for treatment for 12 weeks, then receive GC-MRT for 12 weeks.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Gaze Contingent Music Reward Therapy — Feedback according to participants' viewing patterns, in order to modify their attention.
  Arms: Gaze Contingent Music Reward Therapy
Drug: Escitalopram — 10-20 mg of Escitalopram
  Other Names: Cipralex
  Arms: Selective Serotonin Reuptake Inhibitors
Behavioral: Waitlist — Participants will wait for 12 weeks while in touch with the clinic, then receive GC-MRT for 8 weeks.
  Arms: Waitlist Control

SUMMARY:
The purpose of this study is to determine the clinical efficacy and neuro-cognitive mechanisms of Gaze-Contingent Usic Reward Therapy for social anxiety disorder, compared with treatment with SSRIs or waitlist control.

DETAILED DESCRIPTION:
Attention biases in threat processing have been assigned a prominent role in the etiology and maintenance of anxiety disorders. The purpose of this study is to determine whether giving gaze-contingent feedback is an effective treatment for social anxiety disorder, compared to treatment with SSRI (Escitelopram) and a waitlist control. A secondary purpose is to explore the unique neuro-cognitive mechanisms of this treatment, using eye-tracking, MRI and fMRI measurements. Participants will be assessed using clinical interviews and self-rated questionnaires before, during and after 12 weeks of treatment or wait. Outcome measures will be social anxiety symptoms, as well as dwell time on threat in eye-tracking paradigms tested in previous studies, and BOLD signals in MRI measurements. Neuro-cognitive mechanisms will be explored as potential mediators of clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* A signed consent form
* Men and women between the ages of 18 and 65.
* Meeting a current diagnosis of Social Anxiety Disorder (SP) according to the DSM-IV.
* SP as the primary diagnosis: In cases of co-morbidity, SP will be deemed as the most distressing and clinically significant condition among the co-morbid disorders.
* No current pharmaco-therapy.

Exclusion Criteria:

* A diagnosis of psychotic or bipolar disorders.
* A diagnosis of a neurological disorder (i.e., epilepsy, brain injury).
* Drug or alcohol abuse.
* Any current pharmacological treatment.
* Any current psychotherapeutic treatment.
* Change in treatment during the study.
* Poor judgment capacity (i.e., children under 18 and special populations).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline - the Liebowitz Social Anxiety Scale - Diagnostic Interview scores | 6 weeks into intervention, 1 week after intervention completion
  The LSAS is a 24-item scale, each item corresponding to a situation selected on the basis of clinical experience. Each item is rated on a severity scale ranging from 0 to 3 with regard to the passing week, measuring separately two components of social anxiety, specifically, fear/anxiety and avoidance of social interaction and performance situations. Although the assessor may request and ask for further detail and adjust the rating based on clinical experience, this option is not often exercised, and inter-rater agreement is not considered to be a relevant concern.

SECONDARY OUTCOMES:
Change from baseline - the Social Phobia Inventory scores | At baseline, at weeks 2,4,6,8,10 of the intervention or wait period, 1 week after intervention completion
  This is a 17-item self-report measure of social anxiety evaluating fear, avoidance and physiological discomfort. Each item is rated on scale ranging from 0 to 4 with a possible total score of 68.
Clinical Global Impression | 6 weeks into intervention, 1 week after intervention completion
  A global measure of clinician impression improvement and severity of illness, ranging from 1 to 7.

OTHER OUTCOMES:
Change from baseline - the Patient Health Questionnaire (PHQ)- a measure of depression | at baseline, one week after end of intervention
  Depression levels at pre and posttreatment and their change from baseline were used as moderators for clinical outcome
Change from baseline - viewing patterns on threat-neutral face matrices | at baseline, 6 weeks into intervention and one week after end of intervention
  gaze patterns, and specifically attention allocation to threat, at pre, mid and posttreatment and their change from baseline were used as moderators for clinical outcome, as well as indicators of target engagement for the GCMRT group. This is done using an established eye-tracking task (Lazarov et al, 2016). Data will also be extracted from the training sessions of GC-MRT participants to evaluate change during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azriel O, Arad G, Tik N, Weiser M, Bloch M, Garber E, Lazarov A, Pine DS, Tavor I, Bar-Haim Y. Neural activation changes following attention bias modification treatment or a selective serotonin reuptake inhibitor for social anxiety disorder. Psychol Med. 2024 Sep 10;54(12):1-13. doi: 10.1017/S0033291724001521. Online ahead of print. PMID 39252484
- [Derived] Arad G, Azriel O, Pine DS, Lazarov A, Sol O, Weiser M, Garber E, Bloch M, Bar-Haim Y. Attention Bias Modification Treatment Versus a Selective Serotonin Reuptake Inhibitor Or Waiting List Control for Social Anxiety Disorder: A Randomized Clinical Trial. Am J Psychiatry. 2023 May 1;180(5):357-366. doi: 10.1176/appi.ajp.20220533. Epub 2023 Mar 22. PMID 36945823